CLINICAL TRIAL: NCT07215572
Title: Implementing a Group Physical Therapy Program for Veterans With Knee Osteoarthritis: Function QUERI 3.0 (QUE 25-008)
Brief Title: Implementing a Group Physical Therapy Program for Veterans (GroupPT): Function QUERI 3.0
Acronym: GroupPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 25-002
Record Dates: First submitted 2025-10-06; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Knee Osteoarthritis
Keywords: Veterans; Implementation Science; Functional Status; Physical Therapy; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Parallel cluster-randomized trial (parallel-CRT): used in pragmatic evaluations of health program or policy interventions, where half the clusters (in this case, VA sites) are randomly assigned to two interventions: Foundational support only (active comparator) vs. Foundational support plus Reach+Equity Implementation Bundle (experimental).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Foundational Support (Active Comparator): Foundational Support uses the Replicating Effective Program (REP) implementation strategy and includes 5 elements that were developed and tested in our prior Function QUERI work: shareholder engagement, Group PT toolkit, Online shared resources (SharePoint) access for clinical program training materials, data reports to assist sites with tracking their data, and Diffusion Networks to promote peer-to-peer sharing and implementation support.
  Interventions: Other: Implementation Strategy: Foundational Support
- Reach+Equity Bundle (Experimental): The Reach+Equity bundle will include the same activities as foundational support plus the Reach+Equity bundle activities which include: 1) external facilitation (provide an outside perspective to help sites identify barriers, develop effective strategies, and navigate complex change processes particularly through the lens of achieving equitable reach); 2) equity in implementation toolkit (guide that supports awareness and consideration of health equity during the implementation process); and 3) equity-focused data-driven monitoring (inform progress regarding equitable reach-related goals).
  Interventions: Other: Implementation Strategy: Reach+Equity Bundle

INTERVENTIONS:
Other: Implementation Strategy: Foundational Support — Foundational Support uses the Replicating Effective Program (REP) implementation strategy and includes 5 elements that were developed and tested in our prior Function QUERI work: shareholder engagement, Group PT toolkit, Online shared resources (SharePoint) access for clinical program training materials, data reports to assist sites with tracking their data, and Diffusion Networks to promote peer-to-peer sharing and implementation support.
  Other Names: Foundational REP
  Arms: Foundational Support
Other: Implementation Strategy: Reach+Equity Bundle — The Reach+Equity bundle will include the same activities as foundational support plus the Reach+Equity bundle activities which include: 1) external facilitation (provide an outside perspective to help sites identify barriers, develop effective strategies, and navigate complex change processes particularly through the lens of achieving equitable reach); 2) equity in implementation toolkit (guide that supports awareness and consideration of health equity during the implementation process); and 3) equity-focused data-driven monitoring (inform progress regarding equitable reach-related goals).
  Other Names: Enhanced Support
  Arms: Reach+Equity Bundle

SUMMARY:
Implementing Group Physical Therapy for Veterans with Knee Osteoarthritis (Group PT): Function QUERI 3.0 aims to compare implementation approaches while also gathering information on clinical effects of the EBP in its new context. The overall goal is to address a key priority within the implementation science field - identifying and refining metrics for equity and impact. The overall goal is to implement, evaluate, and sustain GroupPT in 20 VA facilities using a type III effectiveness-implementation hybrid study framework and parallel CRT design.

DETAILED DESCRIPTION:
Background/Purpose. Exercise-based PT is a key component of guideline concordant knee OA management. However, PT is underutilized for knee OA, resulting in missed opportunities to improve outcomes for the many Veterans with this health condition. A key challenge is the high demand for PT services for knee OA, paired with limited availability of PT services, which can lead to long wait times for Veterans or high community care costs for the VA. Group-based delivery of PT for knee OA can enhance access and efficiency. Following the RCT that supported the effectiveness of Group PT relative to individual PT, the Durham Veterans Affairs Healthcare System (DVAHCS) offered Group PT as a clinical service, and found that patients achieved clinically relevant improvements in pain and functional outcomes that were comparable to those observed in the RCT. Most recently, the investigators conducted a 19-site trial comparing implementation strategies to support delivery of Group PT in the VA. Overall, 16 sites successfully delivered a Group PT program, enrolling a total of 366 Veterans. There were clinically relevant improvements in pain interference and functional outcomes among participating Veterans.

Aims:

Aim 1: Refine foundational REP and Reach+Equity to support implementation of Group PT.

Key Questions: How can the Reach+Equity bundle be optimized to facilitate equitable reach? What are shareholder perspectives on refinements needed for Group PT foundational REP activities, as well as strategies to enhance equitable reach (Reach+Equity bundle)? Aim 2: Evaluate implementation of Group PT with foundational REP versus foundational REP and Reach+Equity. Key Questions: Are there differences in implementation outcomes (reach, fidelity, adoption, cost) at six, 12 and 18 months between arms? Is reach representative of patients experiencing knee OA at participating sites (equitable reach) and does this differ between foundational REP and Reach+Equity arms? Are there differences in effectiveness outcomes (function, pain) between arms? How do sites experience implementation strategies in each arm?

Methodology. To evaluate implementation of Group PT (Aim 2), the investigators will randomize sites (n=20) 1:1 to either foundational support or foundational support plus the Reach+Equity bundle. Implementation activities will occur over a 12-month period. Foundational REP will feature an extensive Implementation Toolkit that includes specific guidance for EBP delivery (e.g., flow of the class, specific exercises, didactic content), along with comprehensive patient resources including videos to guide home exercise. The Reach+Equity bundle will include: 1) external facilitation (provide an outside perspective to help sites identify barriers, develop effective strategies, and navigate complex change processes particularly through the lens of achieving equitable reach); 2) equity in implementation toolkit (guide that supports awareness and consideration of health equity during the implementation process); and 3) equity-focused data-driven monitoring (inform progress regarding equitable reach-related goals). The Group PT sessions includes 6 sessions that include exercise and educational content. Patients will be eligible for Group PT if they have a clinician diagnosis of symptomatic knee OA and ineligible if they have a substantial fall risk or co-occurring health conditions that would make participation in a group exercise class unsafe. The primary follow-up outcome time point will be 18 months; metrics will also be evaluated at 6 and 12 months. Implementation outcomes include: Reach (primary), defined as the number of patients initiating Group PT, Fidelity, defined as the average number of sessions attended by patients who initiate the EBP, and Adoption, defined as launching a Group PT program and enrolling 5 Veterans. Effectiveness Outcomes/Quality Metrics will be collected during the Group PT sessions and documented in the electronic health record. These outcomes include the PROMIS Pain Interference and Function scales, a 30-second chair stand test, and patient satisfaction. Generalized linear models will be used to examine the effect of foundational vs. Reach+Equity on reach and fidelity. Generalized linear mixed effect models will be used to compare effective outcomes between implementation arms.

ELIGIBILITY:
Inclusion Criteria:

Sites are eligible to participate if they have:

* 2 outpatient PT clinicians (one primary and one back-up) for delivering Group PT
* space to conduct group sessions (if delivering Group PT in person) or ability to conduct visits via telehealth (video)

Patients will be eligible for Group PT if they have a clinician diagnosis of symptomatic knee OA.

Exclusion Criteria:

* Site will be ineligible to participate if they are already conducting a group physical therapy class for patients with knee OA.
* Patients will be ineligible for Group PT if they have a substantial fall risk or co-occurring health conditions that would make participation in a group exercise class unsafe.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Reach | 18 months
  Reach (primary) will be defined as the number of patients initiating Group PT.

SECONDARY OUTCOMES:
Reach | 6 months
  Reach (primary) will be defined as the number of patients initiating Group PT.
Reach | 12 months
  Reach (primary) will be defined as the number of patients initiating Group PT.
Fidelity | 6 months
  Fidelity will be defined as the average number of sessions attended by patients who initiate the EBP.
Fidelity | 12 months
  Fidelity will be defined as the average number of sessions attended by patients who initiate the EBP.
Fidelity | 18 months
  Fidelity will be defined as the average number of sessions attended by patients who initiate the EBP.
Adoption | 6 months
  Adoption will be defined as launching a Group PT program and enrolling ≥5 Veterans.
Adoption | 12 months
  Adoption will be defined as launching a Group PT program and enrolling ≥5 Veterans.
Adoption | 18 months
  Adoption will be defined as launching a Group PT program and enrolling ≥5 Veterans.

OTHER OUTCOMES:
PROMIS Pain Interference | 6 months
  A self-reported measure that captures the consequences of pain on relevant aspects of life, including engagement with social, cognitive, emotional, physical, and recreational activities. Lower scores are better, indicating less pain interference. The investigators will use the PROMIS v1.1 Pain Interference Short form 4a.
PROMIS Physical Function | 6 months
  A self-reported measure that captures the difficulty of performing instrumental activities of daily living. Higher scores are better, indicating more physical function. The investigators will use the PROMIS Short form 4a PROMIS v2.0 Physical Function Short form 4a.
PROMIS Pain Interference | 12 months
  A self-reported measure that captures the consequences of pain on relevant aspects of life, including engagement with social, cognitive, emotional, physical, and recreational activities. Lower scores are better, indicating less pain interference. The investigators will use the PROMIS v1.1 Pain Interference Short form 4a.
PROMIS Pain Interference | 18 months
  A self-reported measure that captures the consequences of pain on relevant aspects of life, including engagement with social, cognitive, emotional, physical, and recreational activities. Lower scores are better, indicating less pain interference. The investigators will use the PROMIS v1.1 Pain Interference Short form 4a.
PROMIS Physical Function | 12 months
  A self-reported measure that captures the difficulty of performing instrumental activities of daily living. Higher scores are better, indicating more physical function. The investigators will use the PROMIS Short form 4a PROMIS v2.0 Physical Function Short form 4a.
PROMIS Physical Function | 18 months
  A self-reported measure that captures the difficulty of performing instrumental activities of daily living. Higher scores are better, indicating more physical function. The investigators will use the PROMIS Short form 4a PROMIS v2.0 Physical Function Short form 4a.
30-second Chair Stand Test | 6 months
  Number of times patient can stand up from a seated position and sit back down within 30 seconds.
30-second Chair Stand Test | 12 months
  Number of times patient can stand up from a seated position and sit back down within 30 seconds.
30-second Chair Stand Test | 18 months
  Number of times patient can stand up from a seated position and sit back down within 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Dominick Allen, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be available upon request. Prior to distribution, a local privacy officer and study statistician will certify that the dataset contains no protected health information (PHI). Data will be provided to requestor in electronic format. Sufficient data and descriptors will be made available to duplicate statistical analysis and confirm conclusions in publication. No data or statistical code that could lead to re-identification of individuals will be released. Data will be stored & maintained in an approved, secured location as described in the VA Research Data Inventory Form. The statistician will create de-identified, publication-specific datasets that includes variables from statistical models presented in publication. Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re-identify any individual whose data are included in the dataset.
Supporting Information: Study Protocol
Time Frame: Available upon request.
Access Criteria: Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re- identify any individual whose data are included in the dataset.
URL: https://www.durham.hsrd.research.va.gov/Function_Independence_QUERI.asp